CLINICAL TRIAL: NCT03132454
Title: Phase I Study of Palbociclib Alone and in Combination in Patients With Relapsed and Refractory Leukemias
Brief Title: Palbociclib and Sorafenib, Decitabine, or Dexamethasone in Treating Patients With Recurrent or Refractory Leukemia
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0772; NCI-2018-01194 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0772 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-04-25; First posted 2017-04-27 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Recurrent Acute Lymphoblastic Leukemia; Recurrent Acute Myeloid Leukemia; Refractory Acute Lymphoblastic Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute | interventions — Decitabine; Injections; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; palbociclib; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm I (palbociclib, sorafenib) (Experimental): Patients receive palbociclib PO QD on days 1-28. Patients also receive sorafenib PO QD on days 1-28 beginning on cycle 2. Treatment repeats every 28 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Palbociclib; Drug: Sorafenib
- Arm II (palbociclib, decitabine) (Experimental): Patients receive palbociclib as in Arm I. Beginning cycle 2, patients receive palbociclib PO QC on days 1-7 and decitabine IV QD over 1 hour on days 8-17 of cycle 2 and days 8-12 of cycles 3-8. Treatment repeats every 28 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Decitabine; Drug: Palbociclib
- Arm III (palbociclib, dexamethasone) (Experimental): Patients receive palbociclib as in Arm I. Patients also receive dexamethasone PO QD or IV over 15-30 minutes on days 1-4 and 15-18 beginning on cycle 2. Treatment repeats every 28 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dexamethasone; Drug: Palbociclib

INTERVENTIONS:
Drug: Decitabine — Given IV
  Other Names: 5-Aza-2''-deoxycytidine; Dacogen; Decitabine for Injection; Deoxyazacytidine; Dezocitidine
  Arms: Arm II (palbociclib, decitabine)
Drug: Dexamethasone — Given IV or PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
  Arms: Arm III (palbociclib, dexamethasone)
Drug: Palbociclib — Given PO
  Other Names: 6-Acetyl-8-cyclopentyl-5-methyl-2-((5-(piperazin-1-yl)pyridin-2-yl)amino)-8h-pyrido(2,3-d)pyrimidin-7-one; Ibrance; PD 0332991; PD 332991; PD 991; PD-0332991
Drug: Sorafenib — Given PO
  Other Names: BA4 43 9006; BAY 43-9006; Bay-439006
  Arms: Arm I (palbociclib, sorafenib)

SUMMARY:
This phase I trial studies the side effects and best dose of palbociclib when given alone and in combination with sorafenib, decitabine, or dexamethasone in treating patients with leukemia that has come back (recurrent) or that does not respond to previous treatment (refractory). Palbociclib, sorafenib, and decitabine may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as dexamethasone, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving palbociclib alone and in combination with sorafenib, decitabine, or dexamethasone may work better in treating patients with recurrent or refractory leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) and dose limiting toxicities (DLT) of various combinations with palbociclib in patients with relapsed and refractory leukemias.

SECONDARY OBJECTIVES:

I. To assess pharmacodynamic effects of palbociclib on the Cyclin-CDK-Rb axis in leukemic blasts of patients with relapsed/refractory (R/R) leukemias.

II. To explore the efficacy (complete response [CR], complete remission without platelet recovery [CRp], complete remission without blood count recovery [CRi], partial response [PR], or clinical benefit [CB]) of palbociclib as a single-agent and in combinations in patients with R/R leukemias.

III. To explore biomarkers of response and resistance in patients with R/R leukemias treated with palbociclib.

IV. To assess the safety and tolerability of one cycle of single-agent palbociclib in patients with R/R leukemias.

OUTLINE: This is a dose-escalation study of sorafenib, decitabine, and dexamethasone. Patients are assigned to 1 of 3 arms.

ARM I: Patients receive palbociclib orally (PO) once daily (QD) on days 1-28. Patients also receive sorafenib PO QD on days 1-28 beginning on cycle 2. Treatment repeats every 28 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive palbociclib as in Arm I. Beginning cycle 2, patients receive palbociclib PO QC on days 1-7 and decitabine intravenously (IV) QD over 1 hour on days 8-17 of cycle 2 and days 8-12 of cycles 3-8. Treatment repeats every 28 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity.

ARM III: Patients receive palbociclib as in Arm I. Patients also receive dexamethasone PO QD or IV over 15-30 minutes on days 1-4 and 15-18 beginning on cycle 2. Treatment repeats every 28 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with a diagnosis of histologically confirmed relapsed or refractory (R/R) acute myeloid leukemia or R/R acute lymphoblastic leukemia for which no available standard therapies are indicated or anticipated to result in a durable response.
2. Only participants with R/R ALL will be eligible for cohort C
3. Age >/= 15 years.
4. Participants must not have had leukemia therapy for 14 days prior to starting palbociclib. However, participants with rapidly proliferative disease may receive hydroxyurea as needed until 24 hours prior to starting therapy on this protocol and starting the first cycle of study.
5. Adequate organ function as defined below:

   * liver function (bilirubin < 2mg/dL, AST and/or ALT <3 x ULN - or <5 x ULN if related to leukemic involvement)
   * kidney function (creatinine < 1.5 x ULN ).
   * known cardiac ejection fraction of > or = 45% within the past 3 months
6. ECOG performance status of ≤ 2.
7. A negative urine pregnancy test is required within 1 week for all women of childbearing potential prior to enrolling on this trial.
8. Participants must have the ability to understand the requirements of the study and signed informed consent. A signed informed consent by the participants or his legally authorized representative is required prior to their enrollment on the protocol.

Exclusion Criteria:

1. Participants women are excluded from this study because the agent used in this study has the potential for teratogenic or abortifacient effects. Because there is a potential risk for adverse events in nursing infants secondary to treatment of the mother with the chemotherapy agents, breastfeeding should also be avoided.
2. Uncontrolled intercurrent illness including, but not limited to active uncontrolled infection, symptomatic congestive heart failure (NYHA Class III or IV), unstable angina pectoris, clinically significant cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
3. Participant with documented hypersensitivity to any of the components of the therapy program.
4. Participants with active, uncontrolled CNS leukemia will not be eligible.
5. Men and women of childbearing potential who do not practice contraception. Women of childbearing potential and men must agree to use contraception prior to study entry and for the duration of study participation.
6. Participants with known history of serous retinopathy will not be eligible.
7. Prior treatment with palbociclib,

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) as determined by dose limiting toxicity (DLT) | Up to cycle 2 (each cycle is 28 days)
  MTD is defined as the highest dose level in which 6 patients have been treated with at most 1 instance of dose limiting toxicity using a classic '3+3' dose-escalation design. DLT is defined as drug-related adverse events during cycle two (i.e., the first cycle of palbociclib in combination). The number and proportion of DLTs will be summarized by treatment arm and dose level.

SECONDARY OUTCOMES:
Pharmacodynamic (PD) effects of palbociclib | Up to 3 years
  PD biomarker concentration will be summarized by time points. The relationship between drug concentrations and PD effects will be explored graphically. Based on review of these graphs, analyses to describe the relationship may also be performed.
Efficacy as determined by complete response (CR]), complete remission without platelet recovery (CRp), complete remission without blood count recovery (CRi), partial response (PR), or clinical benefit (CB) | Up to 3 years
  For the preliminary efficacy analysis, the study will summarize the number and rate of CR, CRp, CRi and PR by treatment arm and dose level.
Assessment of biomarkers of response and resistance | Up to 3 years
  The study will also explore the biomarkers associated with response or resistance to treatment using descriptive statistics and exploratory graphics.
Incidence of adverse events graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Tapan M Kadia, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org